CLINICAL TRIAL: NCT05437029
Title: A Phase 1b Study to Assess Safety, Tolerability, and Pharmacokinetics of a Multiple Dosing Schedule of Q-Griffithsin Intranasal Spray for Broad-spectrum Coronavirus Prophylaxis: A Study of the PREVENT-CoV Program
Brief Title: Safety, Tolerability, and Pharmacokinetics of Q-Griffithsin Intranasal Spray
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kenneth Palmer (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Kenneth Palmer, Professor, University of Louisville
Organization: University of Louisville (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 22.0224; MCDC2006-010 (Other Grant/Funding Number: U.S. Department of Defense)
Record Dates: First submitted 2022-05-13; First posted 2022-06-29 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: COVID-19 Prevention
Keywords: COVID-19; Q-griffithsin; Nasal Spray; Prophylactic; Corona Virus; SARs CoV 2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Q-Griffithsin Group 1: 3.0 mg daily spray (Experimental): In Group 1, up to 12 participants will receive a dose of 3.0 mg intranasal Q-GRFT administered once daily, as 2 sprays (100 µL/ spray) in each nostril, for 7 days.
  Interventions: Drug: Q-Griffithsin 3.0
- Q-Griffithsin Group 2: two 3.0 mg sprays per day (Experimental): In Group 2, up to 12 participants will be enrolled to receive a total of 6.0 mg intranasal Q-GRFT administered as 3.0 mg twice daily (3.0 mg BID), with 2 sprays (100 µL/ spray) in each nostril approximately every 12 hours, for 7 days.
  Interventions: Drug: Q-Griffithsin 6.0

INTERVENTIONS:
Drug: Q-Griffithsin 3.0 — This is an open-label dose-escalation study to assess the safety, tolerability, and pharmacokinetics (PK) of a multiple dosing schedule of low dose Q GRFT intranasal spray DP
  Other Names: Q-Griffithsin Group 1
  Arms: Q-Griffithsin Group 1: 3.0 mg daily spray
Drug: Q-Griffithsin 6.0 — This is an open-label dose-escalation study to assess the safety, tolerability, and pharmacokinetics (PK) of a multiple dosing schedule of high dose Q GRFT intranasal spray DP
  Other Names: Q-Griffithsin Group 2
  Arms: Q-Griffithsin Group 2: two 3.0 mg sprays per day

SUMMARY:
The purpose of this study is to test the safety of multiple doses of a Q-GRFT nasal spray in healthy volunteers. This Q-GRFT nasal spray is "investigational and not approved by the FDA for general use" and is being developed to prevent the transmission of COVID-19 and other coronaviruses.

DETAILED DESCRIPTION:
This is an open-label dose-escalation study to assess the safety, tolerability, and pharmacokinetics (PK) of a multiple dosing schedule of Q GRFT intranasal spray DP.

Up to 24 healthy participants will be enrolled and assigned to either of 2 groups to receive treatment. In Group 1, up to 12 participants will receive a dose of 3.0 mg intranasal Q-GRFT administered once daily, as 2 sprays (100 µL/ spray) in each nostril, for 7 days. The initial dose will be administered in the clinic by a study clinician. Participants will be taught how to self-administer the study product at the clinic and receive written instructions for at-home self-administration. Subsequent doses will be self-administered either at the clinic or at home. Group 1 participants will undergo PK sampling (nasal and nasopharyngeal fluids) at baseline (enrollment visit), on day 1 (1 hour, 6 hours, and 10 hours after the initial dose), day 2 (24±1 hours after initial dose), day 4 (pre-dose and 1-hour post-dose), day 7 (pre-dose, 1 hour, 6 hours, and 10 hours after the final dose, day 8 (24±1 hours) and day 9 (48±2 hours) following the final dose. Blood for evaluation of systemic exposure will be collected at baseline, day 1 and day 4 (1 hour post-dose), and on day 8, upon dose completion.

In Group 2, up to 12 participants will be enrolled to receive a total of 6.0 mg intranasal Q-GRFT administered as 3.0 mg twice daily (3.0 mg BID), with 2 sprays (100 µL/ spray) in each nostril approximately every 12 hours, for 7 days. Administration of the third dose among Group 2 participants will be delayed to permit obtaining a 24-hour PK timepoint for one completed 6.0 mg BID treatment. The initial dose will be administered in the clinic by a study clinician. Participants will be taught to self-administer the study product at the clinic and receive written instructions for at-home self-administration. Subsequent doses will be self-administered either at the clinic or at home. Participants in this group will undergo PK sampling (nasal and nasopharyngeal fluids) at baseline (enrollment visit), on day 2 (1 hour, 6 hours, and 10 hours after the second dose), day 3 (24±1 hours after the second dose), day 5 (pre-dose after 3 completed doses of 6 mg and 1 hour post-dose), day 8 (pre-dose, 1 hour, 6 hours, and 10 hours after the final dose), day 9 (24±1 hours) and day 10 (48±2hours) following the final dose. Blood for evaluation of systemic exposure will be collected at baseline, on day 2 and day 5 (1 hour post-dose), and on day 9 after the final dose completion.

Safety assessment for both groups will be conducted after 3 days of dosing, upon completion of the final dose, and within 3-4 weeks of dose completion. An optional rectal fluids sampling procedure using a sponge will be performed 1 day after the final dose, to assess for any study product in the gastrointestinal tract. Blood draws for anti-drug antibodies/ immunogenicity assays will be performed at baseline, 24±1 hours after the final dose and 3-4 weeks after the final dose administration. Additional participants will be enrolled in case any subjects do not complete all safety or primary PK assessments, in order to assure that a minimum of 9 subjects is available for full analysis. All sampling procedures will be performed in the clinic.

This sample size is appropriate for a Phase 1b clinical study to gather additional multi-dosing safety data and preliminary PK data following completion of the single-dose treatment Phase 1a trial. The proposed studies will allow a careful selection of the ideal dose that will be administered to subjects in future Phase 2 studies.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 negative using Rapid antigen test at screening.
* Able and willing to provide written informed consent to take part in the study.
* Able and willing to provide adequate information for locator purposes.
* Availability to return for all study visits, barring unforeseen circumstances.
* Agree not to participate in other research studies involving drugs and/or medical devices during the study period.
* Female participants must meet the following criteria:

Postmenopausal or using (or willing to use) an acceptable form of contraception (e.g., barrier method, IUD, hormonal contraception, sexual abstinence, surgical sterilization, or vasectomization of male partner).

If the female participant has female partners only, the method of contraception will be noted as a barrier method for study documentation.

Not be pregnant at the baseline or enrollment visit. Not be breastfeeding at screening or intend to breastfeed during study participation per participant report.

* Willingness and ability to defer vaccinations until after study participation is completed. This does not include COVID-19 vaccinations.
* Participants should have received all COVID-19 vaccines that they are eligible for. Those eligible for booster doses will not delay getting their dose for purposes of enrolling in the study. They will first obtain their booster dose and be re-evaluated for enrollment 2 weeks following their booster dose.
* Willingness to perform at-home study product self-administration according to written instructions that will be provided.
* Willingness to follow local guidelines for mask-wearing and face coverings.
* Must be in general good health in the opinion of the investigator.

Exclusion Criteria:

* Participants with ongoing moderate to severe allergic rhinitis, asthma, or history of chronic obstructive pulmonary disease (COPD), and currently suffering from chronic rhinitis or acute/chronic sinusitis.
* Participants who report any of the following at Screening:

  1. Ongoing common cold or flu-like symptoms for 48 hours prior to the screening, including sore throat, blocked nose, runny nose, cough, and sneezing.
  2. Participants who experience moderate or severe or higher seasonal allergies, such as hay fever, (symptoms in excess of mild, intermittent nasal rhinorrhea, sneezing, or itchy/watery eyes).
  3. Non-therapeutic injection drug use in the 6 months prior to screening and recreational snorting drug use or on prescription medication/ concomitant therapy other than for contraception and antibiotics. Those excluded will include individuals taking prescription medications like systemic steroids, intranasal medicines, among others.
  4. Participants who are current smokers.
  5. Known allergy to methylparaben, or propylparaben, or any ingredients of the formulated drug product.
  6. Use of systemic immunomodulatory medications (Thalidomide, Lenalidomide, Pomalidomide, Imiquimod, etc.), anticoagulants, and other drugs assessed by the site Investigator within the 4 weeks prior to study enrollment.
  7. History of alcohol/ substance abuse within 6 months of study enrollment.
  8. History of any vaccinations within the 2 weeks prior to enrollment.
  9. Participating in another research study involving drugs or medical devices within the 4 weeks prior to enrollment.
  10. Having plans to relocate away from the study site area during the period of study participation.
* Has any of the following laboratory abnormalities at Screening:

  1. White blood cell count < 2,000 cells/mm3 or > 15,000 cells/mm3.
  2. Hemoglobin <12 g/dL for men and <11 g/dL for women.
  3. Calculated creatinine clearance >1.1 x upper limit of normal (ULN).
  4. Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) > 1.1 × the site laboratory ULN.
  5. Total bilirubin > 1.1 x ULN.
  6. ≥ +1 glucose or +2 protein on urinalysis (UA).
* Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study, or unable to comply with the study requirements. Such conditions may include but are not limited to a current or recent history (within last 6 months) of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral disease, severe nasal septum deviation, or other condition that may cause nasal obstruction like nasal polyps or nasal/ sinus surgery in the past.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic levels | Nasopharyngeal fluids on days 1, 2, 4, 7, 8, 9 for group 1; Days 2, 3, 5, 8, 9 for group 2
  Q-GRFT Study Product (SP) concentration will be assessed in nasopharyngeal fluids.
Safety of product by measuring number of subjects that experience Adverse Events greater than Grade 3. | 3-4 weeks
  Incidence of AEs Grade 3 or higher as defined by the Division of AIDS (DAIDS) Table or Grading the Severity of Adult and Pediatric Adverse Events, V2.1 (July 2017).

SECONDARY OUTCOMES:
Smell Assessment by Brief Smell Identification Test | Visit 0, 6 or 7 (Day 9)
  Smell Assessment will be performed using the Sensonics International Brief Smell Identification Test (BSIT) to evaluate the impact of Q GRFT SP intranasal treatment on the sensation. This is a "scratch and sniff" type test with a set number of defined odors that participants should be able to identify. Modification of smell perception can be identified by changes in the results of the BSIT>
Acceptability | 3 - 4 weeks
  The product acceptability will be assessed to determine perception of use by participants. This is achieved through a assessing participants' responses to defined questions on a questionnaire that asks how the participants feel about their experiences with the investigational nasal spray product, and how likely they might be to use the product if it is approved for use. A majority of answers indicating a negative impression of the user experience will alert the study team to the possibility that the product will not be acceptable for use if approved and marketed as a nasal spray to prevent virus infection.
Quality of life outcome | Visit 0, 6 or 7 (Day 9)
  Quality of Life will be evaluated with the SF-12 battery of questions. The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
Anti-drug antibody levels | Day 8 or 9
  Anti-drug antibodies (ADA) will be measured in collected plasma to assess if any anti-QGRFT antibodies are generated after multiple Q-GRFT SP treatment
Pharmacokinetic levels | 3 - 4 weeks
  Q-GRFT Study Product (SP) concentration will be assessed in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald W Dryden, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Clinical Trials Unit, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doty RL, Marcus A, Lee WW. Development of the 12-item Cross-Cultural Smell Identification Test (CC-SIT). Laryngoscope. 1996 Mar;106(3 Pt 1):353-6. doi: 10.1097/00005537-199603000-00021. PMID 8614203
- [Background] Chen H, Cisternas MG, Katz PP, Omachi TA, Trupin L, Yelin EH, Balmes JR, Blanc PD. Evaluating quality of life in patients with asthma and rhinitis: English adaptation of the rhinasthma questionnaire. Ann Allergy Asthma Immunol. 2011 Feb;106(2):110-118.e1. doi: 10.1016/j.anai.2010.10.027. Epub 2011 Jan 8. PMID 21277512
- [Background] Doty RL. Office procedures for quantitative assessment of olfactory function. Am J Rhinol. 2007 Jul-Aug;21(4):460-73. doi: 10.2500/ajr.2007.21.3043. PMID 17882917
- [Derived] Cash E, Deitz K, Potts KL, Nabeta HW, Zahin M, Rai SN, Dryden GW, Palmer KE. Development and validation of a product acceptability questionnaire for intranasal Q-Griffithsin COVID-19 prophylaxis (SPRAY PAL). BMJ Open. 2023 Sep 12;13(9):e073735. doi: 10.1136/bmjopen-2023-073735. PMID 37699630